CLINICAL TRIAL: NCT02327585
Title: Study on the Psychological Behavior Intervention Technology of Attention Deficit Hyperactivity Disorder
Brief Title: Behavioral Intervention for Children With Attention Deficit Hyperactivity Disorder(ADHD)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Min Chen (Other)
Responsible Party: Sponsor-Investigator, Min Chen, postgraduate, Peking University
Organization: Peking University (Other)
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-4024-04
Record Dates: First submitted 2014-12-12; First posted 2014-12-30 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Executive function training; child
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Executive function training (Experimental): Children diagnosis of ADHD are randomized to the experimental condition(Executive Function training) or waiting group experimental:participants will receive 12 sessions of executive function training weekly no intervention :waiting participants will not be treated with executive function therapy and keep waiting for 12 weeks for comparison
  Interventions: Behavioral: A randomized controlled study of Executive Function training for children with ADHD

INTERVENTIONS:
Behavioral: A randomized controlled study of Executive Function training for children with ADHD — Children diagnosis of ADHD are randomized to the experimental condition(Executive Function therapy) or waiting group experimental:participants will receive 12 sessions of executive function therapy weekly no intervention :waiting participants will not be treated with executive function therapy and keep waiting for 12 weeks for comparison

SUMMARY:
ADHD children have executive function (EF) impairments,so we randomize the children to the training or a waitlist to improve EF ,adding contingent reinforcement to ascertain whether EF deficits are amenable to the training in children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of child ADHD
* full-scale intelligence quotient (FSIQ) ≥70
* stable on medication for ADHD children at least 3 months

Exclusion Criteria:

* individuals with major neurological disorders
* a diagnosis of schizophrenia, epilepsy, mental retardation or other brain disorders

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
change in ADHD-rating scale | baseline,after the training (12week)

SECONDARY OUTCOMES:
change in behavior rating scale of executive function | baseline,after the training (12week)
cambridge Neuropsychological Test Automatic Battery | baseline,after the training (12week)
Conners | baseline,after the training (12week)

CONTACTS AND LOCATIONS:
Overall Officials: li yang, PHD MD, Study Director — Peking University
Locations (1):
- Peking University Sixth Hospital/Institute of Mental Health, Beijing, China

REFERENCES:
- [Derived] Qian Y, Chen M, Shuai L, Cao QJ, Yang L, Wang YF. Effect of an Ecological Executive Skill Training Program for School-aged Children with Attention Deficit Hyperactivity Disorder: A Randomized Controlled Clinical Trial. Chin Med J (Engl). 2017 Jul 5;130(13):1513-1520. doi: 10.4103/0366-6999.208236. PMID 28639564